CLINICAL TRIAL: NCT05663502
Title: Biospecimen Collection and Donation to the AIDS and Cancer Specimen Resource (ACSR): A Companion Protocol to AMC Trials
Brief Title: Collecting Blood and Tissue Sample Donations for Research for HIV/AIDS-Related Cancers
Status: Recruiting | Type: Observational
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AMC-S005; NCI-2021-05722 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC-S005 (Other: AIDS Malignancy Consortium); AMC-S005 (Other: CTEP); UM1CA121947 (NIH)
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Anal Carcinoma; Hematopoietic and Lymphoid Cell Neoplasm; HIV Infection; Kaposi Sarcoma; Lymphoma; Malignant Solid Neoplasm; Multicentric Castleman Disease; Plasmablastic Lymphoma; Recurrent Kaposi Sarcoma; Recurrent Lymphoma; Recurrent Plasmablastic Lymphoma; Transplant-Related Kaposi Sarcoma
MeSH Terms: conditions — Anus Neoplasms; Hematologic Neoplasms; HIV Infections; Sarcoma, Kaposi; Lymphoma; Multi-centric Castleman's Disease; Plasmablastic Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational (biospecimen collection): Patients undergo collection of fresh blood and/or tumor tissue samples
  Interventions: Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and/or tumor tissue sample collection
  Other Names: Biological Sample Collection

SUMMARY:
This study collects blood and tissue samples for research of human immunodeficiency virus (HIV)/acquired immunodeficiency syndrome (AIDS)-related cancers. Collecting blood and tissue samples and studying biomarkers in the laboratory may help doctors to learn how are biologic or genetic factors related to HIV and cancers that occur commonly in people living with HIV.

DETAILED DESCRIPTION:
This study is collecting blood and tissue samples (biospecimens) from people living with HIV, who are participating in an AIDS Malignancy Consortium (AMC) clinical trial. Biospecimens are also collected from people who are not living with HIV, but who have a type of cancer that is common in persons living with HIV. The National Cancer Institute created the AIDS and Cancer Specimen Resource (ACSR), a place where these tissue samples are stored, so researchers can learn more about how to treat HIV and related diseases. The AMC works with the AIDS and Cancer Specimen Resource (ACSR) to collect donated samples from people living with HIV or who have cancers that are associated with HIV for future research studies. People who do not take part in an AMC clinical trial can donate samples to the ACSR.

Individuals who agree to participate will be asked to donate blood once. Their blood will be stored in a biobank, and used for research. Individuals may also donate tissue - either from a previous procedure, or from an upcoming procedure.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years of age
* Participant must be HIV- positive and have a diagnosed malignancy. If participants are HIV-negative, they must have a newly diagnosed or recurrent malignancy that has an established scientific connection (e.g., shared etiology) to an AIDS- associated malignancy such as:

  * classic Kaposi sarcoma
  * transplant-associated Kaposi sarcoma,
  * anal cancer,
  * multicentric Castleman's disease,
  * Epstein Barr Virus (EBV) -positive lymphoma
  * plasmablastic lymphoma
  * Hodgkin's lymphoma.

    * For participants that are HIV-positive, HIV infection must be documented by means of any one of the following: :

      * Documentation of HIV diagnosis in the medical record by a licensed health care provider;
      * Documentation of receipt of antiretroviral therapy (ART) by a licensed health care provider (Documentation may be a record of an ART prescription in the participant's medical record, a written prescription in the name of the participant for ART, or pill bottles for ART with a label showing the participant's name. Receipt of at least two agents is required; each component agent of a multi-class combination ART regimen will be counted toward the 2-agent requirement, excepting receipt of a pre-exposure prophylaxis (PrEP) regimen alone [e.g., Truvada], which is exclusionary);
      * HIV ribonucleic acid (RNA) detection by a licensed HIV RNA assay demonstrating > 1000 RNA copies/mL;
      * Any licensed HIV screening antibody and/or HIV antibody/antigen combination assay confirmed by a second licensed HIV assay such as a HIV Western blot confirmation or HIV rapid multispot antibody differentiation assay.
* Participants with HIV infection, regardless of participation in an AMC clinical trial, must have a diagnosis of cancer, cancer or a condition that places them at a higher risk of cancer.
* The investigator determines that the participant (or his/her legally authorized representative [LAR]) has the ability to provide informed consent and the participant or LAR provides written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population includes patients with human immunodeficiency virus (HIV) infection and HIV-associated malignancies, as well as HIV-negative cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2030-08-31 (Estimated); Study Completion 2035-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of biospecimens collected | Through study completion, anticipated to be 10 years
  The number of blood and tissue specimens will be counted.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Bethony, Principal Investigator — AIDS Malignancy Consortium
Locations (8):
- United States (8):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California, San Francisco, San Francisco, California
  - George Washington University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah